CLINICAL TRIAL: NCT03448549
Title: A Prospective Randomized Controlled Trial to Compare Oxaliplatin Combined With S-1 (SOX) Versus Oxaliplatin With Capecitabine (XELOX) as Adjuvant Chemotherapy for Stage III Colorectal Cancer Patients
Brief Title: SOX Versus XELOX as Adjuvant Chemotherapy for Stage III Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking Union Medical College Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Aiwen Wu, M.D. PH.D. Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKUCH-C02
Record Dates: First submitted 2017-06-04; First posted 2018-02-28 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer Stage III; Adjuvant Chemotherapy
Keywords: Tegafur，gimeracil and oteracil potassium; Capecitabine; compliance; quality of life; adverse reaction; disease free survival; overall survival
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance | interventions — Oxaliplatin; potassium oxonate; Capecitabine

STUDY DESIGN:
Intervention Model Description: Patients enrolled are randomized into SOX group and XELOX group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (TGOP-OX) (Experimental): Colorectal cancer patients p-staged III are randomized and assigned with TGOP-OX (Tegafur，gimeracil and oteracil potassium+Oxaliplatin) as adjuvant chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Tegafur，gimeracil and oteracil potassium
- Group B (XELOX) (Active Comparator): Colorectal cancer patients p-staged III are randomized and assigned with XELOX (Xeloda+Oxaliplatin) as adjuvant chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Xeloda

INTERVENTIONS:
Drug: Oxaliplatin — adjuvant chemotherapy
Drug: Tegafur，gimeracil and oteracil potassium — adjuvant chemotherapy
  Arms: Group A (TGOP-OX)
Drug: Xeloda — adjuvant chemotherapy
  Other Names: Capecitabine
  Arms: Group B (XELOX)

SUMMARY:
Fluorouracil combined with oxaliplatin are routinely recommended to patients with pathological stage III (p-stage III) colorectal cancer, leading to significant improvement of 5-year disease-free survival and overall survival (approximately 3.4% -4.2%) by by international guidelines such as the National Cancer Comprehensive Network. The Considerable proportion of patients suffer with hand-foot syndrome due to capecitabine as commonly prescribed. Meanwhile as another agent of fluorouracil, tegafur，gimeracil and oteracil potassium (short for TGOP) has been shown with similar effect and less adverse reaction. This study was designed to investigate the short-term and long-term safety and efficacy of TGOP-OX and XELOX regimens in colorectal cancer p-stage III patients who undergo curative surgery and adjuvant chemotherapy, and to explore the compliance and quality of life in patients treated with TGOP-OX regime.

DETAILED DESCRIPTION:
In patients with pathological stage III colorectal cancer, capecitabine combined with oxaliplatin, as routinely prescribed for adjuvant chemotherapy prolongs the patient's 5-year disease-free survival and overall survival (about 3.4% -4.2%) and is therefore recommended by the National Comprehensive Cancer Network (NCCN), European Society for Medical Oncology (ESMO) and other international guidelines. Accumulating evidence has shown that a majority of chemotherapy-related side effects were caused by capecitabine, especially in certain patients with hand-foot syndrome lasting a long time. Tegafur，gimeracil and oteracil potassium (TGOP), as another fluorouracil, was shown to be equally effective for colorectal cancer patients as adjuvant chemotherapy. The results of two multicenter randomized controlled trials (Adjuvant Chemotherapy Trial of S-1 for Colon Cancer and Adjuvant Chemotherapy Trial of S-1 for RectalCancer) reported at the American Society of Clinical Oncology (ASCO) 2015 suggested that patients with stage III colorectal cancer treated with tegafur，gimeracil and oteracil potassium (TGOP) instead of capecitabine for adjuvant chemotherapy resulted in comparative effects (5 year Disease free survival: 61.7% -70.2%; 5-year Overall survival: 66.4% -86.0%) with significant lower 3/4 degrees of adverse events. As a compound combined with tegafur, gimeracil and oteracil potassium in a molar ratio of 1: 0.4: 1, it plays an anti-tumor effect as 5-Fu precursor drug, metabolized by liver cytochrome enzyme (P450) system into 5-Fu with less toxicity. The addition of tegafur improves the anti-tumor activity by raising its oral absorption. Gimeracil, as a potent and reversible inhibitor of dihydropyrimidine dehydrogenase (DPD enzyme), largely increases the concentration of 5-Fu in blood and tumor tissue, meanwhile reduces the 5-Fu no active metabolite fluoride-β-alanine (F-β-Ala) production, leading to the decrease of cardiovascular and neural toxicity and the incidence of hand-foot syndrome . Oteracil potassium specifically inhibits the intestinal mucosal cells within the orotate phosphoribosyl transferase (OPRT enzyme), blocking 5-Fu phosphorylation, reducing the digestive tract mucosal damage, thereby lowering the digestive tract toxicity.

Colorectal cancer patients who undergo curative surgery, are enrolled in this study, and randomized into TGOP combined with oxaliplatin (TGOP-OX) and capecitabine combined with oxaliplatin (XELOX) groups. The aim of the study is to confirm that the efficacy of TGOP-OX group as adjuvant chemotherapy is not inferior to that of the XELOX group. Adverse reactions will be systemically collected based on CTCAE 4.0 criteria for each cycle. The quality of life was assessed by the European Cancer Research Organization questionnaires. Patients will undergo close follow-up according to the NCCN recommendation. Minimum follow-up period is designed as 3 years, and each endpoint will be evaluated as each check-point.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form;
* age ≥18 years old;
* randomization within 2-8 weeks after surgery;
* Performance status of the US Eastern Cancer Cooperative Group (ECOG) score 0-1;
* pathologically diagnosed as stage III colon or rectal adenocarcinoma patient;
* Accept effective contraceptive measures;
* postmenopausal women; pregnancy test negative 72 hours before randomization;
* R0 resection.

Exclusion Criteria:

* primary tumor metastasis (including tumor cells in the ascites or the occurrence of peritoneal metastasis);
* presence of clinical relevant cardiovascular disease;
* presence of disease history of central nervous system, or evidence confirmed subjects suffering from central nervous system diseases;
* presence of grade 3 (or over grade 3) peripheral neuropathy, according to the common adverse event evaluation criteria (CTCAE) v. 3.0;
* post-operative radiotherapy must be implemented in patients according to researchers' assessment,;
* presence of any unresolved toxicity left from previous anti-cancer treatment left > grade 2 according to CTCAE, except hair loss;
* simultaneous use of targeted therapeutic drugs, such as anti-vascular endothelial growth factor (VEGF) monoclonal antibody, or anti-epidermal growth factor receptor (EGFR) monoclonal antibody;
* brain metastases or meningeal metastases;
* Insufficiency of bone marrow reserve capacity, the presence of neutrophils absolute count ≤ 1.5 × 109 / L or platelet count ≤ 75 × 109 / L, or the need for regular blood transfusion in order to maintain hemoglobin ≥ 9g / dL;
* Serum bilirubin ≥1.5 × upper limit of reference range (ULRR);
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.5 × ULRR;
* serum creatinine ≥ 1.5 × ULRR or Cockcroft-Gault formula calculated creatinine clearance ≤ 50ml / min;
* Evidence of any severe or uncontrolled systemic disease (eg, unstable or decompensated breathing, heart, liver or kidney disease, HIV infection, hypertension, severe arrhythmia, diabetes, massive active bleeding);
* undergo a major surgery within 14 days prior to entering the study, or surgical incision that has not yet healed completely;
* women who are pregnant or breastfeeding, or women who are positive for pregnancy before the trial;
* subjects known to be allergic to oxaliplatin, capecitabine, S-1 or any ingredient of these products;
* combination of other anti-cancer treatment (including gonadotropin-releasing hormone agonists, anti-cancer Chinese medicine, immunotherapy), except for steroid hormones;
* In the past 5 years there are other malignant tumor history, except curative treatment of skin basal cell carcinoma and / or cervical cancer in situ;
* have a significant history of gastrointestinal damage, the researchers judge may significantly affect the absorption of S-1, including dysphagia;
* subjects known suffering dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1191 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
3 year disease free survival | 3 years
  3 year disease free survival

SECONDARY OUTCOMES:
major adverse event -short term | 6 month after randomiztion (period during post-operational chemotherapy)
  short term adverse reaction is defined as the as event within 3 months after chemotherapy,will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
major adverse reaction-long term | upto 24 months
  long term adverse reaction is defined as the as event 3 months after chemotherapy will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
3 year overall survival | 3 years
  3 year overall survival
The accuracy of assessment of preoperative CT images on the stage | within 3 months before surgery
  The accuracy of assessment of preoperative CT images on the stage(T and N)

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No